CLINICAL TRIAL: NCT05880810
Title: Continuous Glucose Monitor Use for Mayo Clinic Advanced Care at Home Patients With Diabetes Mellitus
Brief Title: Continuous Glucose Monitor for Mayo Clinic Advanced Care at Home Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian G. Dumitrascu, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-000733
Record Dates: First submitted 2023-05-16; First posted 2023-05-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
Keywords: Advanced Care at Home Program (home hospital)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous Glucose Monitoring (Experimental): Subjects admitted to the Advanced Care at Home program (home hospital) will have the continuous glucose monitor sensor placed for up to 10 days to monitor and dose insulin.
  Interventions: Device: Continuous Glucose Monitor Dexcom G6 PRO
- Control Arm (Standard of Care) (No Intervention): Subjects admitted to the Advanced Care at Home program (home hospital) will continue with standard of care glucose monitoring (capillary glucose levels checked via glucometer), insulin dosing, and DM treatment during the 10 day period.

INTERVENTIONS:
Device: Continuous Glucose Monitor Dexcom G6 PRO — Connected to a smart phone that transmits continuous glucose monitoring data in real time to Advanced Care at Home Command Center for monitoring.
  Arms: Continuous Glucose Monitoring

SUMMARY:
The purpose of this study is to measure differences in diabetes control with the use of continuous glucose monitor (CGM) and diabetes education compared with standard of care for glucose monitoring (glucometer checks) and diabetes education in participants with diabetes mellitus receiving therapy with insulin and being admitted to Mayo Clinic Advanced Care at Home Program (ACH).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to Advanced Care at Home (ACH) Program and supposed to remain in ACH for at least 72 hours.
* Patients with previous diagnosis of DM type 1 or type 2.
* Patients taking subcutaneous (SQ) insulin either via multidose injections or SQ insulin pump.
* Capable of giving signed informed consent

Exclusion Criteria:

* Actively treated for diabetes ketoacidosis (DKA) or hyperosmolar hyperglycemic state (HHS).
* Participants taking acetaminophen more than 4g per day or more than 1gm every 6 hours.
* Participants with altered mental status.
* Participants diagnosed with dementia.
* Patients with suicidal ideations or experiencing suicidal behavior.
* Patients with liver cirrhosis.
* Patients with End Stage Renal Disease on dialysis bot hemodialysis or peritoneal dialysis.
* Participants with allergy to medical grade adhesive or medical tape.
* Participants taking hydroxyurea.
* Participants who are pregnant, wanting to become pregnant, or nursing during study period.
* Patients with a planned MRI within the following 10 days after admission to ACH.
* Participants currently using continuous glucose monitor (CGM) to dose insulin or check glucose level.
* Participants with diabetes mellitus (DM) treated with diet alone.
* Participants with DM treated with oral hypoglycemic medications.
* Participants with DM treated with one SQ insulin injection daily.
* Participants enrolled in other studies addressing CGM use.
* Participants physically or emotionally incapable of handling a cell phone with a smart display.
* Participants with hearing impaired to a degree that they are not able to hear a smart phone alert or alarm.
* Patients lacking WIFI or Cellular coverage needed to connect the monitoring cell phone to Internet network.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Time in Range | 10 days
  Percentage of time with continuous glucose monitor values within 70-180 mg/dl
Mean daily glucose | 10 days
  Mean daily glucose level (mg/dl)

SECONDARY OUTCOMES:
Frequency of hypoglycemia episodes | 10 days
  Number of episodes with blood glucose below 70 mg/dl measured via point of care testing (POCT) and Continuous Glucose Monitor (CGM)
Mean absolute relative difference (MARD) variation with Oxygen saturation. | 10 days
  Measured in percentage
Mean absolute relative difference (MARD) variation with Daily hemoglobin. | 10 days
  Measured in grams per deciliter (g/dl)
Mean absolute relative difference (MARD) variation with Glomerular filtration rate (GFR) | 10 days
  Measured in ml/min
Mean absolute relative difference (MARD) variation with Arterial blood pressure | 10 days
  Measured in millimeters of mercury (mmHg)
Percentage of subjects to continue use of continuous glucose monitor | 40 days
  Percentage of subjects will using continuous glucose monitor at 40 days post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Dumitrascu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No